CLINICAL TRIAL: NCT04406753
Title: Is it Possible to Improve the Flexion-rotation Test With an Indirect Approach of C0-1 and C2-3 Segments? A Randomized Controlled Trial.
Brief Title: Indirect Approach of C0-1 and C2-3 Segments in Flexion-rotation Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez-Sanz, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N13/2020
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Neck Pain; Cervical Spine Disease; Rotation
Keywords: manual therapy; neck pain; exercise; restriction
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Nucleolin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy + Exercise Group (Experimental): Manual Therapy + Exercise group will carry out 20-minute session of treatment. The techniques will be applied depending on the clinical findings in each patient and the objective will be to restore the function of C0-1 and C2-3 segments before applying cervical exercises. We will use manipulation (high velocity low amplitude) and/or mobilization (low velocity high amplitude) techniques of C0-1 and C2-3 segments with cervical exercise. Manipulations will be in the direction of traction, with the head in a neutral position. A maximum of two trials at each level on each side will perform (2-6 thrusts). Mobilization will be performed for 5 minutes using repeating cycles of 45 seconds of mobilization and 15 seconds of rest. The cervical exercise will perform by this group will follow the same methodology as the Exercise group.
  Interventions: Other: Manual therapy techniques in C0-1 and C2-3 with cervical exercise
- Exercise Group (Active Comparator): This group will perform the cervical stabilization exercise. They will be teach to perform the contraction of deep neck flexor muscle activity with the help of the Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) in supine. Exercise will be always carry out without pain, because pain can be an inhibitor of muscle contraction.
  The Exercise group will carry out one 20-minute session, composed of 2 sets of 10 repetitions, holding each repetition for 10 seconds, a 40-second rest between each repetition and 2 minutes between sets.
  Interventions: Other: Cervical Exercise

INTERVENTIONS:
Other: Manual therapy techniques in C0-1 and C2-3 with cervical exercise — Manual Therapy + Exercise group will carry out 20-minute session of treatment. The techniques will be applied depending on the clinical findings in each patient and the objective will be to restore the function of C0-1 and C2-3 segments before applying cervical exercises. We will use manipulation (high velocity low amplitude) and/or mobilization (low velocity high amplitude) techniques of C0-1 and C2-3 segments with cervical exercise. Manipulations will be in the direction of traction, with the head in a neutral position. A maximum of two trials at each level on each side will perform (2-6 thrusts). Mobilization will be performed for 5 minutes using repeating cycles of 45 seconds of mobilization and 15 seconds of rest. The cervical exercise will perform by this group will follow the same methodology as the Exercise group.
  Arms: Manual Therapy + Exercise Group
Other: Cervical Exercise — This group will perform the cervical stabilization exercise. They will be teach to perform the contraction of deep neck flexor muscle activity with the help of the Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) in supine. Exercise will be always carry out without pain, because pain can be an inhibitor of muscle contraction.
  The Exercise group will carry out one 20-minute session, composed of 2 sets of 10 repetitions, holding each repetition for 10 seconds, a 40-second rest between each repetition and 2 minutes between sets.
  Arms: Exercise Group

SUMMARY:
Restrictions on upper cervical spine are associated with cervical pain. The vast majority of upper cervical spine rotation occurs at the C1-2 segment. Flexion-rotation test is a valid measure that predominantly measures rotation in C1-2 segment, however upper cervical spine rotation also implies C0-1 and C2-3 due to ligament anatomy. Restriction in flexion-rotation may be due to direct restriction in C1-2, but also to a premature tightening of the alar ligament as a result of lack of movement in C0-1 or C2-3.

The objective is to compare the effect of a 20-minutes single cervical exercise session with or without manual therapy of C0-1 and C2-3 segment in flexion-rotation test in patients with chronic neck pain and positive flexion-rotation test.

To carry out the objective, the following will be designed a randomized controlled assessor-blind clinical trial with primary healthcare patients.

This population will be patients with chronic neck pain and positive flexion-rotation test. These patients will be assigned in manual therapy + exercise group or in exercise group.

Exercise will be focused on deep anterior cervical muscles. Manual therapy will combine techniques in C0-1 and C2-3 with this exercise. Flexion-rotation test, neck pain intensity, pain intensity during the flexion-rotation test and cervical range of motion will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* A medical diagnosis of chronic neck pain with more than 3 months of evolution.
* A positive result in the flexion-rotation test (less than 33º or a difference of 10º or more between the two rotations).
* Being over 18 years old.
* Having signed the informed consent.

Exclusion Criteria:

* Contraindications for manual therapy or exercise.
* Having participated in exercise or manual therapy programs in the last three months.
* Presenting warning signs or having suffered a relevant neck trauma.
* An inability to maintain supine position.
* The use of pacemakers (the magnets in the CROM device could alter their signal)
* An inability to perform flexion-rotation test
* Language difficulties.
* Pending litigation or lawsuits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Flexion-rotation test | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  This test is used to see the amount of movement of the upper cervical spine and is the test most used in the literature. It is positive when there is a decrease of 10 degrees or more in the cervical rotation with maximum flexion, in a sense with respect to the contralateral or presents hypomobility of segment C1 with a mobility less than 33º

SECONDARY OUTCOMES:
Neck pain intensity with Numeric Pain Rating Scale | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  The Numeric Pain Rating Scale (NPRS) is a one-dimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes.
Pain intensity during the flexion-rotation test with Numeric Pain Rating Scale | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  It will be recorded if the patient has pain during the flexion-rotation test
Cervical range of motion | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain